CLINICAL TRIAL: NCT03026257
Title: Clinical Assessment of a Regimen of AIR OPTIX® Plus HYDRAGLYDE® Silicone Hydrogel Lenses and HYDRAGLYDE® Containing Lens Care Solutions
Brief Title: Clinical Assessment of a HYDRAGLYDE® Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCW773-P001
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Refractive Errors; Myopia; Hypermetropia
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AOHG (Experimental): Lotrafilcon B contact lenses with added wetting agent, worn bilaterally (in both eyes) for 30 days in a daily wear modality and cared for with either a hydrogen peroxide-based contact lens solution with added wetting agent or a POLYQUAD/ALDOX-preserved contact lens solution with added wetting agent, as randomized
  Interventions: Device: Lotrafilcon B contact lenses with added wetting agent; Device: POLYQUAD/ALDOX-preserved contact lens solution with added wetting agent; Device: Hydrogen peroxide-based contact lens solution with added wetting agent
- Habitual (Active Comparator): Habitual silicone hydrogel contact lenses worn bilaterally for 30 days in a daily wear modality and cared for with participant's habitual multi-purpose solution (MPS)
  Interventions: Device: Samfilcon A contact lenses; Device: Senofilcon C contact lenses; Device: Senofilcon A contact lenses; Device: Comfilcon A contact lenses; Device: Habitual Multi-Purpose Solution (HMPS)

INTERVENTIONS:
Device: Lotrafilcon B contact lenses with added wetting agent — Silicone hydrogel contact lenses
  Other Names: AIR OPTIX® plus HYDRAGLYDE® (AOHG)
  Arms: AOHG
Device: Samfilcon A contact lenses — Habitual silicone hydrogel contact lenses
  Other Names: Bausch + Lomb ULTRA™ (Ultra)
  Arms: Habitual
Device: POLYQUAD/ALDOX-preserved contact lens solution with added wetting agent — Multi-purpose disinfecting solution for contact lens care
  Other Names: OPTI-FREE® PureMoist® (OFPM)
  Arms: AOHG
Device: Hydrogen peroxide-based contact lens solution with added wetting agent — Solution for contact lens cleaning and disinfecting
  Other Names: CLEAR CARE® PLUS/AOSEPT® PLUS with HYDRAGLYDE® (CCP)
  Arms: AOHG
Device: Senofilcon C contact lenses — Habitual silicone hydrogel contact lenses
  Other Names: Johnson & Johnson ACUVUE® VITA™ (Vita)
  Arms: Habitual
Device: Senofilcon A contact lenses — Habitual silicone hydrogel contact lenses with a replacement pair issued after 2 weeks
  Other Names: Johnson & Johnson ACUVUE® OASYS® 2- Week with HYDRACLEAR® PLUS (Oasys)
  Arms: Habitual
Device: Comfilcon A contact lenses — Habitual silicone hydrogel contact lenses
  Other Names: CooperVision® Biofinity® (Biofinity)
  Arms: Habitual
Device: Habitual Multi-Purpose Solution (HMPS) — Multi-purpose solution for contact lens care according to participant's habitual brand, used per manufacturer's instructions
  Arms: Habitual

SUMMARY:
The purpose of this study is to evaluate worn AIR OPTIX® plus HYDRAGLYDE® (AOHG) lenses cleaned and disinfected with HYDRAGLYDE® containing lens solutions compared to each of the control habitual silicone hydrogel (SiHy) lenses cleaned and disinfected with habitual multi-purpose solution (MPS) for cholesterol uptake.

ELIGIBILITY:
Inclusion Criteria:

* Must sign informed consent document;
* Vision correctable to 0.1 (LogMAR) or better in each eye at distance with habitual lenses;
* Manifest cylinder (at screening) less than or equal to 0.75 diopter (D) in each eye and spectacle add <+0.50 D in each eye;
* Current full-time wearer of spherical samfilcon A, comfilcon A, senofilcon C monthly or senofilcon A 2-week replacement lens within the power range of lens powers available;
* Current user of an MPS (excluding OFPM) to care for lenses;
* Willing to answer text messages on a daily basis during the study;
* Willing to discontinue artificial tears during the study and rewetting drops on the days of study visits;
* Use of digital devices (eg, smart phone, tablet, laptop or desktop computer) for 20 consecutive minutes at least twice a week and willing to continue for the duration of the study;
* Other protocol specific inclusion criteria may apply.

Exclusion Criteria:

* Habitual lens wear in an extended wear modality (routinely sleeping in lenses overnight for 1 or more nights per week);
* Any anterior segment infection, inflammation, disease or abnormality that contraindicates contact lens wear;
* History of herpetic keratitis, corneal surgery or irregular cornea;
* Prior refractive surgery;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator;
* Currently using or have not discontinued Restasis®, Xiidra™ and/or topical steroids within the past 7 days;
* Use of mechanical eyelid therapy or eyelid scrubs within 14 days before Visit 1 and not willing to discontinue during the study;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Known pregnancy or lactating;
* Other protocol specific exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Global Med Affairs, GCRA, Study Director — Alcon, A Novartis Division
Locations (8):
- United States (5):
  - Alcon Investigative Site, Birmingham, Alabama
  - Alcon Investigative Site, Cleveland, Ohio
  - Alcon Investigative Site, Columbus, Ohio
  - Alcon Investigative Site, Memphis, Tennessee
  - Alcon Investigative Site, Houston, Texas
- Alcon Investigative Site, Waterloo, Ontario, Canada
- Germany (2):
  - Alcon Investigative Site, Hildesheim
  - Alcon Investigative Site, Jena

REFERENCES:
- [Derived] Shows A, Redfern RL, Sickenberger W, Fogt JS, Schulze M, Lievens C, Szczotka-Flynn L, Schwarz S, Tichenor AA, Marx S, Lemp-Hull JM. Lipid Analysis on Block Copolymer-containing Packaging Solution and Lens Care Regimens: A Randomized Clinical Trial. Optom Vis Sci. 2020 Aug;97(8):565-572. doi: 10.1097/OPX.0000000000001553. PMID 32769842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 study centers located in the United States (5), Germany (2), and Canada (1).
Pre-assignment Details: Of the 323 enrolled, 66 subjects exited as screen failures prior to randomization. An additional 5 subjects were randomized but discontinued prior to treatment. This reporting group includes all randomized and exposed subjects (252). Subject distribution in As Randomized and As Treatment differs due to 3 subjects with lens/solution misallocations.
Groups:
- AOHG/CCP: Lotrafilcon B contact lenses with added wetting agent, worn bilaterally (in both eyes) for 30 days in a daily wear modality and cared for with a hydrogen peroxide-based contact lens solution with added wetting agent
- AOHG/OFPM: Lotrafilcon B contact lenses with added wetting agent, worn bilaterally for 30 days in a daily wear modality and cared for with a POLYQUAD/ALDOX-preserved contact lens solution with added wetting agent
- Biofinity/HMPS: Habitual silicone hydrogel (SiHy) contact lenses worn bilaterally for 30 days in a daily wear modality and cared for with participant's habitual multi-purpose solution (MPS)
- Vita/HMPS; Ultra/HMPS: Habitual SiHy contact lenses worn bilaterally for 30 days in a daily wear modality and cared for with participant's habitual MPS
- Oasys/HMPS: Habitual SiHy contact lenses worn bilaterally for 30 days (replaced after 15 days) in a daily wear modality and cared for with participant's habitual MPS
Period: Overall Study
Arm/Group | AOHG/CCP | AOHG/OFPM | Biofinity/HMPS | Vita/HMPS | Ultra/HMPS | Oasys/HMPS
Started (Randomized and treated, as randomized) | 60 | 64 | 34 | 25 | 23 | 46
Treated (Randomized and treated, as treated) | 58 | 65 | 35 | 24 | 23 | 47
Completed | 54 | 63 | 34 | 24 | 22 | 46
Not Completed | 6 | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and exposed to a study lens on Day 1 or a study regimen (lens and lens care system (LCS)) thereafter (Full Analysis Set).
Groups:
- AOHG/CCP: Lotrafilcon B contact lenses with added wetting agent, worn bilaterally for 30 days in a daily wear modality and cared for with a hydrogen peroxide-based contact lens solution with added wetting agent
- Biofinity/HMPS; Vita/HMPS; Ultra/HMPS: Habitual SiHy contact lenses worn bilaterally for 30 days in a daily wear modality and cared for with participant's habitual MPS
- Total: Total of all reporting groups
Arm/Group | AOHG/CCP | AOHG/OFPM | Biofinity/HMPS | Vita/HMPS | Ultra/HMPS | Oasys/HMPS | Total
Number analyzed (Participants) | 60 | 64 | 34 | 25 | 23 | 46 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (7.0) | 27.8 (6.0) | 28.2 (5.9) | 28.2 (5.7) | 28.8 (7.2) | 30.4 (8.2) | 28.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 49 | 22 | 17 | 17 | 35 | 179
  Male | 21 | 15 | 12 | 8 | 6 | 11 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 1 | 1 | 1 | 3 | 12
  Not Hispanic or Latino | 54 | 62 | 33 | 24 | 22 | 43 | 238
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Ex Vivo Total Cholesterol Uptake at Day 30
Description: The contact lens worn in the right eye was removed and stored dry and frozen until analysis. Total cholesterol uptake (cholesterol and cholesterol esters) was evaluated from a sample of the right contact lenses from each site and measured in micrograms. Lower total cholesterol uptake indicates increased lens performance.
Time Frame: Day 30
Population: Full Analysis Set with cholesterol uptake measured
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | AOHG/CCP | AOHG/OFPM | Biofinity/HMPS | Vita/HMPS | Ultra/HMPS | Oasys/HMPS
Number analyzed (Participants) | 23 | 25 | 24 | 23 | 20 | 28
μg | 0.28 (0.18) | 0.28 (0.48) | 2.17 (1.47) | 4.18 (3.25) | 2.07 (1.48) | 2.19 (2.69)
Statistical Analysis 1: Comparison: AOHG/CCP vs Biofinity/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 2: Comparison: AOHG/CCP vs Vita/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 3: Comparison: AOHG/CCP vs Ultra/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 4: Comparison: AOHG/CCP vs Oasys/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 5: Comparison: AOHG/OFPM vs Biofinity/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 6: Comparison: AOHG/OFPM vs Vita/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 7: Comparison: AOHG/OFPM vs Ultra/HMPS; Test type: Superiority; p < 0.0001, General Linear Model
Statistical Analysis 8: Comparison: AOHG/OFPM vs Oasys/HMPS; Test type: Superiority; p < 0.0001, General Linear Model

ADVERSE EVENTS:
Time Frame: Lens insertion (Day 1) through study completion, an average of 30 days
Description: Adverse events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. This analysis population includes all subjects/eyes exposed to study lens and/or study LCS evaluated in this study as a regimen (Safety Analysis Set). "At risk" population for ocular AEs is reported in units of eyes, as treated.
Groups:
- AOHG/CCP Ocular: Eyes exposed to AOHG contact lenses and CCP for lens care
- AOHG/CCP Nonocular: Subjects exposed to AOHG contact lenses and CCP for lens care
- AOHG/OFPM Ocular: Eyes exposed to AOHG contact lenses and OFPM for lens care
- AOHG/OFPM Nonocular: Subjects exposed to AOHG contact lenses and OFPM for lens care
- Habitual SiHy/MPS Ocular: Eyes exposed to habitual SiHy contact lenses and habitual MPS for lens care
- Habitual SiHy/MPS Nonocular: Subjects exposed to habitual SiHy contact lenses and habitual MPS for lens care
Arm/Group | AOHG/CCP Ocular | AOHG/CCP Nonocular | AOHG/OFPM Ocular | AOHG/OFPM Nonocular | Habitual SiHy/MPS Ocular | Habitual SiHy/MPS Nonocular
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/58 | 0/130 | 0/65 | 0/258 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/58 | 0/130 | 0/65 | 0/258 | 0/129
Other Adverse Events (participants affected / at risk) | 0/116 | 0/58 | 0/130 | 0/65 | 0/258 | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03026257/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03026257/SAP_001.pdf